CLINICAL TRIAL: NCT01513291
Title: A Phase IIa, Multicenter, Randomized, Placebo-Controlled Clinical Trial to Evaluate the Safety and Efficacy of MK-6096 for Migraine Prophylaxis in Patients With Episodic Migraine
Brief Title: A Study of the Safety and Efficacy of MK-6096 for Migraine Prophylaxis in Participants With Episodic Migraine (MK-6096-020)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 6096-020
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Results first posted 2016-07-20 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Migraine; Headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — MK-6096

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MK-6096 (Experimental): Participants were randomized to receive double-blind MK-6096, two 5 mg tablets (10 mg dose), orally, once daily for 12 weeks in the Treatment Period. Those who completed the Treatment Period were randomized 1:1 to receive double-blind MK-6096 or placebo once daily in the 2-week Run-out Period.
  Interventions: Drug: MK-6096; Drug: Placebo
- Placebo (Placebo Comparator): Participants were randomized to receive double-blind placebo, two tablets, orally, once daily for 12 weeks in the Treatment Period. Those who completed the Treatment Period continued to receive double-blind placebo once daily in the 2-week Run-out Period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-6096 — MK-6096, two 5 mg tablets (total 10 mg dose), orally, once daily
  Arms: MK-6096
Drug: Placebo — Placebo, 2 tablets, orally, once daily

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of MK-6096 versus placebo for preventing migraines in participants with episodic migraine. After a 28-day Screening period during which baseline number of monthly migraine days was assessed, participants were randomized to receive MK-6096 or placebo for a 12-week Treatment Period. Participants who completed all 12 weeks of the Treatment Period received drug or placebo for an additional 2 weeks in the Run-out Period. Treatment assignment in the Run-out Period was determined at the initial randomization. In the Run-out Period, participants who received placebo in the Treatment Period continued to receive placebo and participants who received MK-6096 in the Treatment Period 2 received either MK-6096 or placebo in a 1:1 ratio. The hypothesis tested in the study is that MK-6096 10 mg is superior to placebo in reducing migraine frequency as measured by the mean change from baseline in monthly migraine days averaged over the 12- week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* History of migraine with or without aura for >1 year and with ≥4 and ≤14 migraine days per month in the 3 months prior to study
* Male, female not of reproductive potential, or female of reproductive potential who is not pregnant by pregnancy test and agrees to use acceptable contraception

Exclusion Criteria:

* Pregnancy, breast-feeding, or expecting to become pregnant
* Planning to donate egg or sperm during the study or within 90 days after last dose of study medication
* Basilar or hemiplegic migraine headache
* >50 years old at the age of migraine onset
* ≥15 headache-days per month or medication taken for acute migraine or other headaches on more than 10 days per month in any of the three months prior to study
* Migraine prophylactic medication (defined as medication taken daily to prevent migraines) taken in the 30 days prior to study
* History of narcolepsy, cataplexy, circadian rhythm disorder, parasomnia, sleep related breathing disorder, restless legs syndrome, periodic limb movement disorder, excessive daytime sleepiness or difficulty sleeping due to a medical condition (e.g., asthma, gastroesophageal reflux disease, etc.)
* Clinical, laboratory, or electrocardiogram (ECG) evidence of uncontrolled hypertension, uncontrolled diabetes, human immunodeficiency virus (HIV) disease, or significant pulmonary, renal, hepatic, endocrine, or other systemic disease
* Myocardial infarction, unstable angina, coronary artery bypass surgery, or other revascularization procedure, stroke, or transient ischemic attack within 3 months of study
* Other confounding pain syndromes (i.e., condition requiring daily use of opioids), psychiatric conditions such as uncontrolled major depression, dementia or significant neurological disorders other than migraine
* Imminent risk of self-harm, based on clinical interview and responses on the Columbia Suicidality Severity Rating Scale (C-SSRS), or of harm to others. Exclude any prospective participant reporting suicidal ideation with intent, with or without a plan in the past 2 months or suicidal behavior in the past 6 months
* History of malignancy ≤5 years prior to study, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* History of hypersensitivity to more than two chemical classes of drugs, including prescription and over-the-counter medications
* Recent history (within the past 1 year) or current evidence of drug or alcohol abuse or "recreational use" of illicit drugs or prescription medications
* Donated blood products or has had phlebotomy of >300 ml within 8 weeks of study, or intends to donate blood products or receive blood products within 30 days before study and throughout study
* Consumption of 3 or more alcoholic drinks per day
* Body Mass Index >40 kg/m^2
* History of transmeridian travel (across >3 time zones) or shift work (defined as permanent night shift or rotating day/night shift work) within the past 2 weeks or anticipates needing to travel (across >3 time zones) at any time during the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 237 (Actual)
Dates: Start 2012-02-06 (Actual); Primary Completion 2012-10-03 (Actual); Study Completion 2012-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Chabi A, Zhang Y, Jackson S, Cady R, Lines C, Herring WJ, Connor KM, Michelson D. Randomized controlled trial of the orexin receptor antagonist filorexant for migraine prophylaxis. Cephalalgia. 2015 Apr;35(5):379-88. doi: 10.1177/0333102414544979. Epub 2014 Aug 8. PMID 25106663

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 423 participants were screened. Of these, 237 participants completed screening and met the eligibility criteria, including the required number of migraine days during the Screening period.
Groups:
- Treatment Period: MK-6096: Participants received double-blind MK-6096, two 5 mg tablets (10 mg dose), orally, once daily for 12 weeks in the Treatment Period
- Treatment Period: Placebo: Participants received double-blind placebo, two tablets, orally, once daily for 12 weeks in the Treatment Period
- Run-out Period: MK-6096 / MK-6096: Participants who received MK-6096 and completed the Treatment Period, and were randomized to receive double-blind MK-6096, two 5 mg tablets (10 mg dose), orally, once daily for 2 weeks in the Run-out Period.
- Run-out Period: MK-6096 / Placebo: Participants who received MK-6096 and completed the Treatment Period, and were randomized to receive double-blind placebo, two tablets, orally, once daily for 2 weeks in the Run-out Period.
- Run-out Period: Placebo / Placebo: Participants who received placebo and completed the Treatment Period, received double-blind placebo, two tablets, orally, once daily for 2 weeks in the Run-out Period.
Period: Treatment Period
Arm/Group | Treatment Period: MK-6096 | Treatment Period: Placebo | Run-out Period: MK-6096 / MK-6096 | Run-out Period: MK-6096 / Placebo | Run-out Period: Placebo / Placebo
Started | 120 | 117 | 0 | 0 | 0
Treated | 120 | 115 | 0 | 0 | 0
Completed | 97 | 101 | 0 | 0 | 0
Not Completed | 23 | 16 | 0 | 0 | 0
Not completed — Adverse Event | 8 | 4 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 3 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 5 | 0 | 0 | 0
Not completed — Randomized not treated | 0 | 2 | 0 | 0 | 0
Period: Run-out Period
Arm/Group | Treatment Period: MK-6096 | Treatment Period: Placebo | Run-out Period: MK-6096 / MK-6096 | Run-out Period: MK-6096 / Placebo | Run-out Period: Placebo / Placebo
Started | 0 | 0 | 50 (These participants were pre-randomized from participants in the Treatment Period: MK-6096 group) | 47 (These participants were pre-randomized from participants in the Treatment Period: MK-6096 group) | 101 (These participants were completers from the Treatment Period: Placebo group)
Completed | 0 | 0 | 50 | 45 | 101
Not Completed | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Period: MK-6096 | Treatment Period: Placebo | Total
Number analyzed (Participants) | 120 | 117 | 237
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.5 (10.7) | 41.9 (11.3) | 42.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 99 | 201
  Male | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Monthly Migraine Days
Description: Participants recorded data in the electronic migraine headache diary in the evening approximately one hour before bed and prior to taking study medication during Screening and the Treatment Period. A migraine was defined as a headache with at least one associated symptom of aura, photophobia, phonophobia, nausea, or vomiting. Change in the mean monthly migraine days during Screening (Baseline) versus during the 12-week Treatment Period was assessed. A negative number indicates a reduction in mean monthly migraine days.
Time Frame: Baseline and average over Treatment Period (Weeks 0-12)
Population: The population analyzed included participants who received at least one dose of double-blind study treatment and had at least one evaluable endpoint measurement, including those with only a baseline measurement. This outcome measure applied only to the Treatment Period and was not analyzed for the Run-out Period.
Measure: Least Squares Mean (Standard Error); unit: Days/month
Arm/Group | Treatment Period: MK-6096 | Treatment Period: Placebo
Number analyzed (Participants) | 120 | 114
Days/month
  Baseline | 8.2 (0.1) | 8.2 (0.1)
  Change from Baseline | -1.7 (0.3) | -1.3 (0.3)
Statistical Analysis 1: Comparison: Treatment Period: MK-6096 vs Treatment Period: Placebo; Test type: Superiority or Other; p = 0.33153, Constrained Longitudinal Analysis (cLDA); Risk Difference (RD) = -0.4, 95% CI 2-sided [-1.3 to 0.4] — Risk difference is for MK-6096 - Placebo. The cLDA model included terms for treatment, time, treatment-by-time interaction, monthly migraine days during the Screening (Baseline) Period (≤8, >8) as covariates

2. Primary Outcome: Percentage of Participants With One or More Adverse Events
Description: An adverse event was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the sponsor's product, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the sponsor's product, is also an adverse event. Statistical analysis compared the Treatment Period arms only.
Time Frame: Treatment Period: Weeks 0-12; Run-out Period: Weeks 13-14
Population: The population analyzed included all randomized participants who received at least one dose of double-blind study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Period: MK-6096 | Treatment Period: Placebo | Run-out Period: MK-6096 / MK-6096 | Run-out Period: MK-6096 / Placebo | Run-out Period: Placebo / Placebo
Number analyzed (Participants) | 120 | 115 | 50 | 47 | 101
Percentage of participants | 46.7 | 37.4 | 10.0 | 17.0 | 7.9
Statistical Analysis 1: Comparison: Treatment Period: MK-6096 vs Treatment Period: Placebo; Test type: Superiority or Other; Risk Difference (RD) = 9.3, 95% CI 2-sided [-3.4 to 21.6] — Risk difference (MK-6096 - Placebo) was estimated based on the Miettinen & Nurminen method

3. Primary Outcome: Percentage of Participants Discontinued From Study Medication Due to an Adverse Event
Description: as for outcome 2
Time Frame: Treatment Period: Weeks 0-12; Run-out Period: Weeks 13-14
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Period: MK-6096 | Treatment Period: Placebo | Run-out Period: MK-6096 / MK-6096 | Run-out Period: MK-6096 / Placebo | Run-out Period: Placebo / Placebo
Number analyzed (Participants) | 120 | 115 | 50 | 47 | 101
Percentage of participants | 6.7 | 4.3 | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Treatment Period: MK-6096 vs Treatment Period: Placebo; Test type: Superiority or Other; Risk Difference (RD) = 2.3, 95% CI 2-sided [-4.0 to 8.9] — Risk difference (MK-6096 - Placebo) was estimated based on the Miettinen & Nurminen method

4. Secondary Outcome: Mean Change From Baseline in Monthly Headache Days
Description: Participants recorded data in the electronic migraine headache diary in the evening approximately one hour before bed and prior to taking study medication during Screening and the Treatment Period. A headache was defined as headache pain of at least 30 minutes duration or for any duration for which headache treatment was administered. Change in the mean monthly headache days during Screening (Baseline) versus during the 12-week Treatment Period was assessed. A negative number indicates a reduction in mean monthly headache days.
Time Frame: Baseline and average over Treatment Period (Weeks 0-12)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Days/month
Arm/Group | Treatment Period: MK-6096 | Treatment Period: Placebo
Number analyzed (Participants) | 120 | 114
Days/month
  Baseline | 9.6 (0.2) | 9.6 (0.2)
  Change from Baseline | -1.7 (0.3) | -1.2 (0.3)
Statistical Analysis 1: Comparison: Treatment Period: MK-6096 vs Treatment Period: Placebo; Test type: Superiority or Other; p = 0.24008, Constrained Longitudinal Analysis (cLDA); Risk Difference (RD) = -0.5, 95% CI 2-sided [-1.4 to 0.4] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction From Baseline in Monthly Migraine Days
Description: Participants recorded data in the electronic migraine headache diary in the evening approximately one hour before bed and prior to taking study medication during Screening and the Treatment Period. A migraine was defined as a headache with at least one associated symptom of aura, photophobia, phonophobia, nausea, or vomiting. Percentage of participants with at least 50% reduction in the monthly migraine days during the 12-week Treatment Period versus during Screening (Baseline) was analyzed using a generalized linear mixed effects model.
Time Frame: Baseline and average over Treatment Period (Weeks 0-12)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment Period: MK-6096 | Treatment Period: Placebo
Number analyzed (Participants) | 115 | 112
Percentage of participants | 24.7 (0.3) [18.8 to 31.6] | 21.1 (0.3) [15.7 to 27.8]
Statistical Analysis 1: Comparison: Treatment Period: MK-6096 vs Treatment Period: Placebo; Test type: Superiority or Other; p = 0.43093, Generalized linear mixed effects model; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.7 to 2.0] — Odds ratio is for MK-6096 / Placebo. The generalized linear mixed effects model included terms for treatment, time, treatment-by-time interaction, monthly migraine days during the Screening (Baseline) Period 1 (≤8, >8) as covariates

6. Secondary Outcome: Percentage of Participants With at Least a 30% Reduction From Baseline in Monthly Migraine Days
Description: Participants recorded data in the electronic migraine headache diary in the evening approximately one hour before bed and prior to taking study medication during Screening and the Treatment Period. A migraine was defined as a headache with at least one associated symptom of aura, photophobia, phonophobia, nausea, or vomiting. Percentage of participants with at least 30% reduction in the monthly migraine days during Screening (Baseline) versus during the 12-week Treatment Period was analyzed using a generalized linear mixed effects model.
Time Frame: Baseline and average over Treatment Period (Weeks 0-12)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment Period: MK-6096 | Treatment Period: Placebo
Number analyzed (Participants) | 115 | 112
Percentage of participants | 40.7 (0.3) [33.7 to 48.1] | 40.5 (0.3) [33.5 to 48.0]
Statistical Analysis 1: Comparison: Treatment Period: MK-6096 vs Treatment Period: Placebo; Test type: Superiority or Other; p = 0.97370, Generalized linear mixed effects model; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.7 to 1.5] — Odds ratio is for MK-6096 / Placebo. The generalized linear mixed effects model included terms for treatment, time, treatment-by-time interaction, monthly migraine days during the Treatment Period 1 (≤8, >8) as covariates

ADVERSE EVENTS:
Time Frame: Treatment Period: Weeks 0-12; Run-out Period: Weeks 13-14.
Description: All Patients as Treated included all randomized participants who received at least one dose of double-blind study treatment.
Groups:
- Run-out Period: Placebo / Placebo: Participants who received placebo and completed the Treatment Period, and were randomized to receive double-blind placebo, two tablets, orally, once daily for 2 weeks in the Run-out Period.
Arm/Group | Treatment Period: MK-6096 | Treatment Period: Placebo | Run-out Period: MK-6096 / MK-6096 | Run-out Period: MK-6096 / Placebo | Run-out Period: Placebo / Placebo
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/115 | 0/50 | 0/47 | 0/101
Other Adverse Events (participants affected / at risk) | 26/120 | 10/115 | 1/50 | 4/47 | 1/101
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period: MK-6096 (N=120) | Treatment Period: Placebo (N=115) | Run-out Period: MK-6096 / MK-6096 (N=50) | Run-out Period: MK-6096 / Placebo (N=47) | Run-out Period: Placebo / Placebo (N=101)
Fatigue (General disorders) | 10 (10) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 16 (18) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.